CLINICAL TRIAL: NCT06430736
Title: Prospective Comparison Between Prophylactic and On-demand Use of Tocilizumab in CAR-T Recipients - a Randomized, Two Arm, Open-label, Single-center Trial
Brief Title: PRONTO Trial (PRophylactic Versus ON-demand Use of TOcilizumab)
Acronym: PRONTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRONTO
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Myeloma; Lymphoma; Leukemia
Keywords: Tocilizumab; Myeloma; Leukemia; Lymphoma; CRS; ICANS
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma; Leukemia | interventions — Abortion, Legal

STUDY DESIGN:
Intervention Model Description: Randomized, two arm, open-label, single-center trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab prophylactic (Experimental): In the experimental arm, patients will receive a single standard dose of Tocilizumab (Actemra®) 8 mg/kg b.w. intravenously infused over 1 hour in 250 ml NaCl 0.9%, with completion of the infusion 1 hour prior to the infusion of the CAR-T cells. Prior to Tocilizumab administration, no specific premedication is given. The treatment of eventual subsequent CRS will be identical as in patients in the standard arm.
  Interventions: Drug: Tocilizumab before CAR-T cell infusion
- Tocilizumab on demand (Active Comparator): In the standard arm, patients will receive conventional antipyretics and Tocilizumab at first clinical signs (being grade 1 or higher) of emerging CRS. Tocilizumab will be given at the standard-dose of 8 mg/kg b.w. intravenously over one hour in 250 ml NaCl 0.9%, and it will be repeated after 8 hours for a maximum of four administrations in patients with ongoing signs of CRS. Prior to Tocilizumab administration, no specific premedication is given.
  Interventions: Drug: Tocilizumab at emerging CRS

INTERVENTIONS:
Drug: Tocilizumab before CAR-T cell infusion — Tocilizumab will be given at the standard-dose of 8 mg/kg b.w. intravenously, with completion of the infusion 1 hour prior to infusion of CAR-T cells.
  Treatment of eventual subsequent CRS/ICANS will be identical as in patients in the standard arm.
  Other Names: Prophylactic
  Arms: Tocilizumab prophylactic
Drug: Tocilizumab at emerging CRS — Tocilizumab will be given at the standard-dose of 8 mg/kg b.w. intravenously, and it will be repeated after 8 hours for a maximum of four administrations in patients with ongoing signs of CRS.
  Other Names: On demand
  Arms: Tocilizumab on demand

SUMMARY:
Despite the consequent use of Tocilizumab together with conventional antipyretics at early/first signs of emerging CRS, CRS (and eventually the subsequent development of ICANS) remain a major concern for patients.

This study aims to identify safety and efficacy of prophylactic Tocilizumab treatment. In particular, to explore whether prophylactic Tocilizumab treatment can decrease the incidence and severity of CRS (and subsequent eventual neurotoxicity) following CAR-T-treatment.

DETAILED DESCRIPTION:
Adoptive immunotherapy with CD19 (cluster of differentiation antigen 19) targeting chimeric antigen-receptor (CAR-)T cells is an effective therapeutic strategy against relapsed or refractory B-cell malignancies, including B-cell lymphomas, B-ALL (acute lymphoblastic leukemia) and myeloma. Currently, up to 50 commercial CAR-T-cell treatments are performed annually at the Inselspital in Bern, making it by far the largest center for CAR-T cell treatment in Switzerland.

CAR-T treatment is associated with well-described acute adverse events, including cytokine release syndrome (CRS) and neurotoxicity, termed immune effector cell associated neurologic syndrome (ICANS). CRS (at all grades) occurs in between 42 to 93% of all patients with variations among available products, and ICANS can occur (at all grades) in 21% up to 64%.

Acute complications of CAR-T cell therapy are the result of rapid CAR-T cell expansion and of a hyper-inflammatory state related to cell activation. Interleukin (IL-6) is a central mediator of cytokine-responses in CRS and ICANS together with other cytokines and chemokines involved. IL-6 interacts with its receptor (IL-6R) in either membrane-bound form, leading to "classic" IL-6 signaling after interacting with GP130, or soluble in plasma, where the IL-6 / IL-6R complex interacts with GP130 expressing cells in "trans" IL-6 signaling.

Tocilizumab is a humanized monoclonal antibody that binds the IL-6R in both its soluble and membrane-bound forms. Tocilizumab treatment has become the standard of care for patients presenting with CRS (at all grades), together with antipyretic treatment (grades 1 or 2 at the regular ward) or with vasoactive and/or ventilation support at the intensive care unit (grades 3 and 4).

The study aims to assess the incidence of CRS of all grades, as well as the incidence of ICANS of all grades, the duration of hospitalisation and the need of platelet and erythrocyte transfusion within the first three months after CAR-T treatment in patients receiving prophylactic Tocilizumab compared to patients receiving on-demand Tocilizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to receive commercial CAR-T treatment for all registered indications comprising lymphomas, leukemias or myeloma at a single academic center (Bern Inselspital)
* With written informed consent
* Considered by the investigator to be clinically fit for this treatment
* Patients aged ≥18 years

Exclusion Criteria:

* Previous Tocilizumab treatment within 3 months prior to CAR-T infusion
* Patients with treatment with an investigational compound within 8 weeks prior to CAR-T infusion
* Women who are pregnant or breast feeding, or women intending to become pregnant during the study period; or participants lacking safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases during study treatment and for a total of 12 months; Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of CRS of all grades | 30 days
  Number of patients with CRS of any grade according to the ASTCT (American Society for Transplantation and Cellular Therapy ) Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells ; including use of antipyretics

SECONDARY OUTCOMES:
Incidence of ICANS of all grades | 30 days
  Number of patients with ICANS of any grade according to the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells ; including use of antipyretics
Hospitalization duration | 30 days
  Number of days from admission to discharge from hospital
Erythrocyte transfusion needs | 90 days
  Number of transfusion (erythrocyte) given
Platelet transfusion needs | 90 days
  Number of transfusion (platelet) given
Incidence of admissions to the intensive care unit | 30 days
  Number of admissions to the intensive care unit
Incidence of infections | 90 days
  Number of infections per patient
Overall survival rates | 180 days
  Overall survival assessment are based on physician's reporting of the assessments of the various disease types involved at day 90 and day 180
Progression-free survival rates | 180 days
  Relapse assessment are based on physician's reporting of the assessments of the various disease types involved at day 90 and day 180
IL-6 to monitor CRS | 180 days
  daily assessment of IL-6 during the hospitalisation and at day 90 and day 180
Peripheral molecular CAR-T levels | 180 days
  Peripheral molecular DNA CAR-T level measurement performed at day 0, day 8 and once a month during months 2 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof., Study Chair — Insel Gruppe AG Bern Switzerland
Locations (1):
- Insel Gruppe AG, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months
Access Criteria: email contact: thomas.pabst@insel.ch